CLINICAL TRIAL: NCT04347785
Title: Preoperative, Intraoperative and Postoperative Predictors of Post-clamping Neurologic Deficits During Carotid Endarterectomy With Regional Anesthesia
Brief Title: Predictors of Post-clamping Neurologic Deficits During Carotid Endarterectomy With Regional Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Universidade do Porto (Other)
Responsible Party: Principal Investigator, João Rocha Neves, Consultant of Angiology and Vascular Surgery, MD/MSc, MPH epidemiology, FEBVS, Universidade do Porto
Other Study IDs: 248-18
Record Dates: First submitted 2020-03-26; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Carotid Endarterectomy
Keywords: Carotid Stenosis; regional anesthesia
MeSH Terms: conditions — Carotid Stenosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurologic deficit: All consecutive patients from a tertiary referral center who underwent CEA for carotid artery stenosis who presented alterations in the neurologic examination after ICA clamping during CEA area selected
  Interventions: Procedure: carotid endarterectomy
- control: The control patients are submitted to the same procedure but with no neurologic alterations, are consecutively selected. a 1 to 1 ratio is used
  Interventions: Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: carotid endarterectomy — shunt

SUMMARY:
Patients undergoing carotid endarterectomy may suffer from neurologic deficits (ND) during the carotid cross-clamping due to cerebral hypoperfusion. An associated risk of postoperative stroke incidence is also well established.

The aim of this study is to evaluate the predictive factors associated with ND during CEA performed with RA. The perioperative implications of the ND were also evaluated.

DETAILED DESCRIPTION:
Patients undergoing carotid endarterectomy may suffer from neurologic deficits (ND) during the carotid cross-clamping due to cerebral hypoperfusion. An associated risk of postoperative stroke incidence is also well established.

The aim of this study is to evaluate the predictive factors associated with ND during CEA performed with RA. The perioperative implications of the ND were also evaluated.

All consecutive patients from a tertiary referral center who underwent CEA for carotid artery stenosis (CS) and consecutive patients who presented alterations in the neurologic examination after ICA clamping during CEA are selected. The control patients, submitted to the same procedure but with no neurologic alterations, are consecutively selected.

ELIGIBILITY:
Inclusion Criteria:

* carotid endarterectomy under regional anesthesia
* Postclamping carotid deficit

Exclusion Criteria:

* carotid stenting

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-clamping deficits were defined as any persistent alteration at neurologic examination during the CACC and resistant to hemodynamic adjustment
Sampling Method: Non-Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Stroke | up to 5 years
  An episode of neurological dysfunction caused by focal cerebral, spinal, or retinal infarction.

SECONDARY OUTCOMES:
Clavien-Dindo Classification >3 | 30 days
  Postoperative event life threatining and requiring surgical, endoscopic or radiological intervention

OTHER OUTCOMES:
Major adverse cardiosvascular and cerebrovascular events | up to 5 years
  AMI, Stroke, AHF hospitalization, MALE, MACE, All-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Medicina da Universidade do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
after ethics and data manager authorization

REFERENCES:
- [Result] Pereira-Macedo J, Rocha-Neves JP, Dias-Neto MF, Andrade JPV. Prognostic effect of troponin elevation in patients undergoing carotid endarterectomy with regional anesthesia - A prospective study. Int J Surg. 2019 Nov;71:66-71. doi: 10.1016/j.ijsu.2019.09.015. Epub 2019 Sep 19. PMID 31542388
- [Result] Vieira-Andrade JD, Rocha-Neves JP, Macedo JP, Dias-Neto MF. Onset of Neurological Deficit During Carotid Clamping With Carotid Endarterectomy Under Regional Anesthesia Is Not a Predictor of Carotid Restenosis. Ann Vasc Surg. 2019 Nov;61:193-202. doi: 10.1016/j.avsg.2019.05.025. Epub 2019 Aug 2. PMID 31382007
- [Derived] Pereira-Macedo J, Duarte-Gamas L, Pereira-Neves A, de Andrade JJP, Rocha-Neves J. Short-term outcomes after selective shunt during carotid endarterectomy: a propensity score matching analysis. Neurocirugia (Engl Ed). 2024 Mar-Apr;35(2):71-78. doi: 10.1016/j.neucie.2023.07.006. Epub 2023 Sep 9. PMID 37696419

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT04347785/SAP_000.pdf